CLINICAL TRIAL: NCT01032239
Title: A Randomized, Controlled, Open-label, Parallel-group, Multi-center Study to Compare the Effect of Intrathecal Baclofen Therapy Versus Best Medical Treatment on Severe Spasticity in Post-stroke Patients After 6 Months Active Treatment
Brief Title: SISTERS: Spasticity In Stroke Study - Randomized Study
Acronym: SISTERS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.02.7001
Record Dates: First submitted 2009-12-07; First posted 2009-12-15 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Severe Spasticity
Keywords: Severe spasticity in post-stroke patients
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ITB therapy (Active Comparator): Intrathecal Baclofen therapy (Intrathecal baclofen + implantable pump)
  Interventions: Drug: intrathecal baclofen
- Best Medical Treatment (BMT) (No Intervention): Use one or a combination oral antispastic medication.

INTERVENTIONS:
Drug: intrathecal baclofen — ITB test, implant, 6 months follow-up
  Arms: ITB therapy

SUMMARY:
To demonstrate that Intrathecal Baclofen (ITB) Therapy, compared to Best Medical Treatment (BMT), has superior efficacy in the treatment of severe spasticity in adult post-stroke patients with generalized spastic hypertonia who have not reached their therapy goal with other treatment interventions assessed by a decrease in the average Ashworth Scale (AS) score in the lower extremities.

DETAILED DESCRIPTION:
This is a randomized, controlled open-label parallel group study to demonstrate the efficacy benefit of ITB Therapy over BMT in post-stroke patients with severe spasticity who have not reached their therapy goal with other treatment interventions.

In order to evaluate the efficacy benefit of ITB Therapy over BMT in post-stroke patients, a two-arm parallel group design will be applied. Patients will be equally randomized to one of two treatment arms:

1. ITB Therapy arm; or
2. BMT arm

The study consists of a run-in phase of 21 days for the BMT treatment arm and 2-25 days for the ITB Therapy treatment arm, followed by a 6 month active trial.

The BMT treatment arm will receive a combination of oral antispastic medication and physiotherapy. Patients must be prescribed at least one or a combination of the following oral antispastic medications: oral baclofen, tizanidine, diazepam (or other benzodiazepines) or dantrolene. Following the run-in phase, patients will enter the 6 month active trial.

The ITB Therapy treatment arm will receive a combination of ITB Therapy and physiotherapy. During the run-in phase, a test with intrathecal baclofen will be performed to evaluate the response of the patient. Patients fulfilling the test success criterium will be implanted with a Medtronic SynchroMed®II infusion system. Following implant, patients will enter into the 6 month active trial, which includes a 6 week titration phase, during which time oral antispastic medications must be gradually reduced with complete discontinuation by the end of the titration period.

During the 6 month active trial, patients will be assessed at 3 and 6 months. All primary and secondary endpoint assessments will be performed by a blinded assessor.

The total study duration is expected to be 60 months, including a 39 month enrollment period. The total duration per patient is approximately 7 months (approximately 1 month run-in period followed by 6 months active treatment).

ELIGIBILITY:
Inclusion criteria:

To be eligible for inclusion into this study, patients must fulfill all of the following criteria prior to study enrollment:

1. patient (or legal guardian) has been informed of the study procedures and has given written informed consent
2. patient experienced last stroke > 6 months prior to enrollment
3. patient presents spasticity in at least 2 extremities
4. patient presents an Ashworth score ≥ 3 in a minimum of two of the affected muscle groups in the lower extremities
5. patient is eligible to receive ITB Therapy following the Adult Spasticity Algorithm. A patient does not reach his/her therapy goal with other treatment interventions
6. stable blood pressure: no change in hypertensive medication in last month (NOTE: ventriculoperitoneal shunts and valves can be present)
7. if female, she must either be post-menopausal or surgically sterilized; or use a hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study
8. patient/family is willing to comply with study protocol including attending the study visits

Exclusion criteria:

To be eligible for inclusion in this study the patients must not meet any of the following criteria:

1. patient/family is considered by the physician to be unable or unwilling to participate in long-term ITB Therapy management
2. patient has known hypersensitivity to baclofen
3. active systemic infection (NOTE: pressure sores are not a contraindication unless they are present near the implant sites)
4. presence of a cardiac pacemaker, ICD, implantable neurostimulator or drug delivery device
5. uncontrolled refractory epilepsy
6. use of oral vitamin K antagonists, e.g. warfarin/coumadin; unless the patient can switch to another accepted anticoagulant (e.g. heparin, aggrenox, fragmin, plavix, ticlid) for the period of ITB test and implant
7. patient is pregnant or breastfeeding
8. patient received a Botulinum toxin injection less than 4 months ago

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopold SALTUARI, Prof., Principal Investigator — Landeskrankenhaus Hochzirl, Zirl (Austria)
Locations (25):
- United States (9):
  - University of California Irvine, Irvine, California
  - MedStar National Rehabilitation Network, Washington D.C., District of Columbia
  - Design Neuroscience Center, Doral, Florida
  - Rehabilitation Medical Group - Florida Hospital, Orlando, Florida
  - Tallahassee Neurological Clinic Department of Neurosurgery, Tallahassee, Florida
  - Saint Alphonsus Regional Med Center, Boise, Idaho
  - Research Medical Center, Kansas City, Missouri
  - Einstein Hospital/Moss Rehabilitation, Elkins Park, Pennsylvania
  - TIRR Memorial Herman Hospital, Houston, Texas
- Austria (2):
  - Sozialmedizinisches Zentrum Baumgartner Höhe Otto-Wagner-Spital, Vienna
  - Landeskrankenhaus Hochzirl, Zirl
- Belgium (3):
  - Clin. Univ. UCL Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, campus Pellenberg, Leuven
- Germany (4):
  - Kliniken Beelitz GmbH Neurologische Rehabilitationsklinik, Beelitz-Heilstätten
  - Ambulantes Neurologisches Rehabilitationszentrum, Bonn
  - Therapiezentrum Burgau, Burgau
  - Rhein-Sieg-Klinik Dr. Becker Klinikgesellschaft, Nümbrecht
- Italy (2):
  - Centro di Riabilitazione "Villa Beretta", Costa Masnaga
  - Fondazione Salvatore Maugeri Clinica del lavoro e della riabilitazione IRCSS, Pavia
- Afdeling Revalidatie Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Univerzitetni rehabilitacijski inštitut Republike Slovenije Soča, Ljubljana, Slovenia
- Spain (2):
  - Fundació Privada Institut de Neurorehabilitació Guttmann, Badalona, Barcelona
  - Hospital Universitario La Paz, Madrid
- St George's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Creamer M, Cloud G, Kossmehl P, Yochelson M, Francisco GE, Ward AB, Wissel J, Zampolini M, Abouihia A, Calabrese A, Saltuari L. Effect of Intrathecal Baclofen on Pain and Quality of Life in Poststroke Spasticity. Stroke. 2018 Sep;49(9):2129-2137. doi: 10.1161/STROKEAHA.118.022255. PMID 30354975
- [Derived] Creamer M, Cloud G, Kossmehl P, Yochelson M, Francisco GE, Ward AB, Wissel J, Zampolini M, Abouihia A, Berthuy N, Calabrese A, Loven M, Saltuari L. Intrathecal baclofen therapy versus conventional medical management for severe poststroke spasticity: results from a multicentre, randomised, controlled, open-label trial (SISTERS). J Neurol Neurosurg Psychiatry. 2018 Jun;89(6):642-650. doi: 10.1136/jnnp-2017-317021. Epub 2018 Jan 11. PMID 29326296

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 61 patients were enrolled. One patient did not meet the inclusion criteria (screening failure). 60 patients were then randomized into the study.
Period: Overall Study
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Started | 31 (randomized to ITB arm) | 29 (randomized to BMT arm)
Implant | 25 (implanted) | 0
Completed | 24 | 24
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ITB Therapy | Best Medical Treatment (BMT) | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.09 (11.12) | 55.67 (8.60) | 55.89 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 24 | 18 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 23 | 46
  Other | 8 | 6 | 14
Time since stroke [Mean (Standard Deviation); unit: years] | 4.95 (3.56) | 4.55 (3.73) | 4.76 (3.62)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Ashworth Scale (AS) in Affected Lower Extremities From Baseline to Month 6
Description: AS is a manual test, measuring the resistance to passive movement about a joint with varying degrees of velocity. Scores range from 1-5, with 5 choices. A score of 1 indicates no resistance, and 5 indicates rigidity. The following muscle groups in the lower extremities were assessed: hip flexors, hip adductors, knee extensors, knee flexors, plantar flexors and ankle-dorsal flexors. Average AS was calculated as the average of AS scores of the 6 muscles of the affected lower extremity. Change in average AS in affected lower extremities from baseline to month 6 between ITB and BMT arm was assessed.
  Change= AS at month 6 - AS at baseline.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 25 | 26
units on a scale | -0.99 (0.75) | -0.43 (0.72)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); To test the null hypothesis the sample size needed was 44 evaluable patient (22 per arm) with a power of 80 %; Test type: Superiority; p = 0.0140, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -0.667, 95.1% CI 2-sided [-1.000 to -0.1667]

2. Secondary Outcome: Change in Average Ashworth Scale (AS) in Affected Upper Extremities From Baseline to Month 6
Description: AS is a manual test, measuring the resistance to passive movement about a joint with varying degrees of velocity. Scores range from 1-5, with 5 choices. A score of 1 indicates no resistance, and 5 indicates rigidity. The following muscle groups in the upper extremities were assessed: wrist flexors, elbow flexors, elbow extensors, shoulder abductors and shoulder adductors. Average AS was calculated as the average of AS scores of the 5 muscles of the affected lower extremities. Change in average AS in affected upper extremities from baseline to month 6 between ITB and BMT arm was assessed.
  Change= AS at month 6 - AS at baseline.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 25 | 26
units on a scale | -0.66 (0.59) | -0.17 (0.70)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Test type: Superiority; p = 0.0042, Wilcoxon (Mann-Whitney); Hodges-Lehmann = -0.600, 95% CI 2-sided [-1.0000 to -0.2000]

3. Secondary Outcome: Change in Functional Independence Measure (FIM) Score From Baseline to Month 6
Description: FIM contains 18 items composed of 13 motor tasks and 5 cognitive tasks. Tasks are rated on a 7-point ordinal scale that ranges from total assistance (or complete dependence) to complete independence. Ratings should reflect actual observed performance, not capability. Total score ranges from 18 (lowest) to 126 (highest) level of independence. Change in FIM total score from baseline to month 6 between ITB and BMT arm was assessed. Change=FIM score at month 6 - FIM score at baseline.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 25 | 26
units on a scale | 2.68 (10.31) | -2.58 (11.00)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Test type: Superiority; p = 0.0540, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Average 10 Meter Time Walking Test (10MTWT) From Baseline to Month 6
Description: Change in average 10MTWT from baseline to month 6 beetween ITB and BMT arm. Change=10MTWT at month 6 - 10MTWT at baseline
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.Only High level functional patients (HLP) were analyzed. HLP were defined as patients able to transfer from the wheelchair to bed without human assistance.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 19 | 21
seconds | 4.86 (59.82) | -2.48 (65.60)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Test type: Superiority; p = 0.6256, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants Who Were Able to Transfer From the Wheelchair to Bed Without Human Assistance
Description: Patient was asked to transfer from the wheelchair to bed without human assistance. High level functional patient (HLP) could transfer. Low level functional patient (LLP) was not able to transfer. Comparison of the number and percentage of HLP and LLP between ITB and BMT arms was evaluated.
Time Frame: baseline, month 3, month 6
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 31 | 29
Participants
  Baseline: HLP | 22 | 24
  Baseline: LLP | 9 | 5
  Month 3: number analyzed (Participants) | 25 | 26
  Month 3: HLP | 19 | 21
  Month 3: LLP | 6 | 5
  Month 6: number analyzed (Participants) | 24 | 24
  Month 6: HLP | 19 | 19
  Month 6: LLP | 5 | 5
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Test type: Superiority; p = 0.3676, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change in Numeric Pain Rating Scale (NPRS) From Baseline to Month 6
Description: NPRS is designed to assess the level of pain a patient is feeling at a point in time. The following questions has been presented to patients: What is your actual spasticity-related or spasm-related pain? What was your least spasticity-related or spasm-related pain during the last week? What was your worst spasticity-related or spasm-related pain during the last week? The patient indicated how much pain he is feeling on a scale from 0 to 10. A score of 0 (zero) is "no pain" while a score of 10 (ten) is "worst possible pain". Change in NPRS related to actual, least or worst pain from baseline to month 6 between ITB and BMT arm was assessed. Change=NPRS at month 6 - NPRS at baseline.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 23 | 25
units on a scale
  Actual pain | -1.17 (3.17) | 0.00 (3.29)
  Least Pain | -1.61 (2.29) | 0.24 (3.07)
  Worst Pain | -1.35 (2.42) | -0.04 (3.69)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Actual Pain; Test type: Superiority; p = 0.0380, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Least Pain; Test type: Superiority; p = 0.0136, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Worst Pain; Test type: Superiority; p = 0.2427, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Participants Who Achieved Their Primary Therapeutic Goal Assessed With the Goal Attainment Scale (GAS)
Description: GAS is designed to measure the achievement of treatment goals using the following 6 levels of achievement: worse than start (-3), much less than expected (-2), somewhat less than expected (-1), as expected (0), somewhat more than expected (+1), much more than expected (+2). The primary therapy goal and the criteria for the levels of achievement was defined by the medical team together with the patient and his/her family/legal representative/caregiver at the first day of the study. The number and percentage of patients who achieved the therapeutic goal at Month 6 was compared between the ITB and BMT arm.
Time Frame: month 6
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 24 | 24
Participants
  goal achieved | 10 | 8
  goal not achieved | 14 | 16
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Test type: Superiority; p = 0.7661, Fisher Exact

8. Secondary Outcome: Change in Euro QoL Group-5 Dimensional, 3 Level Version (EQ-5D-3L) From Baseline to Month 6
Description: The EQ-5D-3L is a generic measure of health status consisting in the EQ-5D-3L descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system is characterized on five dimensions: mobility, self-care, ability to undertake usual activities, pain and anxiety/depression. Patients were asked to indicate their level of health on each dimension using one of three levels: "no health problems", "moderate health problems", and "severe health problems". Responses from the questionnaire were converted to a single health index utility score; this ranges from -0.595 to 1. EQ VAS records the patient's self-rated health on a vertical visual analogue scale from 0 to 100 where the endpoints are labelled 'Best imaginable health state' (100) and 'Worst imaginable health state' (0). Change in EQ-5D-3L utility score and VAS score from baseline to month 6 between ITB and BMT arm were assessed. Change=EQ-5D-3L utility or VAS score at month 6 - EQ-5D-3L utility or VAS score.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 25 | 25
units on a scale
  Utility Score | 0.09 (0.26) | 0.01 (0.16)
  VAS | 9.68 (20.42) | 4.40 (21.75)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Utility Score; Test type: Superiority; p = 0.0197, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ITB Therapy vs Best Medical Treatment (BMT); VAS; Test type: Superiority; p = 0.3807, t-test, 2 sided

9. Secondary Outcome: Change in SF-12 (12-item Short Form) From Baseline to Month 6
Description: The SF-12 is generic assessment of health-related quality of life, which evaluates 8 health dimensions (physical functioning, role physical, bodily pain, vitality, social functioning, role emotional, mental health, and general health). Subscale scores for each dimension were aggregated into summary scores for physical (PCS) and mental health (MCS) components (ranging from 0 to 100, with higher scores indicating better health). Changes in the PCS and MCS from baseline to Month 6 were both compared between the BMT and ITB arms. Change=SF-12 score at month 6 - SF-12 score at baseline.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
  SF-12 assessment has been introduced later in a second version of the protocol, hence the lower number of patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 9 | 9
units on a scale
  PCS | 3.13 (3.47) | -1.13 (6.63)
  MCS | 1.05 (10.92) | -0.82 (7.81)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); PCS; Test type: Superiority; p = 0.1068, t-test, 2 sided
Statistical Analysis 2: Comparison: ITB Therapy vs Best Medical Treatment (BMT); MCS; Test type: Superiority; p = 0.6824, t-test, 2 sided

10. Secondary Outcome: Change in Stroke Specific Quality of Life (SS-QoL ) From Baseline to Month 6
Description: SS-QoL questionnaire is a self-assessed quality of life questionnaire specifically designed for post-stroke patients. It evaluates 49 items across 12-domains: personality, energy, language, mobility, vision, upper extremity function, thinking, mood, work/productivity, self-care, and family and social roles. Each item is rated on a 5-point Likert Scale, measuring either positive or negative response to a statement. Summary score is composed of an unweighted average of the 12 domain scores, with higher scores indicating better QoL. Total score ranges from 1 to 5. Change in SS-QoL summary score from baseline to month 6 between ITB and BMT arm was assessed.
  Change=SS-QoL score at month 6 - SS-QoL score at baseline.
Time Frame: Baseline and month 6
Population: Intent to treat analysis. Last Observation Carried Forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 24 | 25
units on a scale | 0.26 (0.58) | 0.05 (0.58)
Statistical Analysis 1: Comparison: ITB Therapy vs Best Medical Treatment (BMT); Test type: Superiority; p = 0.2105, t-test, 2 sided

11. Secondary Outcome: Therapy Satisfaction
Description: Patients were presented with two statements ("I am satisfied with the reduction in spasticity provided by my treatment", and "I would recommend this therapy to a friend"). They agreed, disagreed or were neutral with the statements.
Time Frame: month 6
Population: Intent to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 22 | 23
Participants
  Patient Satisfaction with Spasticity Reduction: disagree | 2 | 7
  Patient Satisfaction with Spasticity Reduction: neutral | 4 | 5
  Patient Satisfaction with Spasticity Reduction: agree | 16 | 11
  Patient Therapy Reccomandation: disagree | 3 | 5
  Patient Therapy Reccomandation: neutral | 3 | 4
  Patient Therapy Reccomandation: agree | 16 | 14

12. Secondary Outcome: Healthcare Resource Utilization
Description: Number of patients with healthcare professional contacts outside of study visits in the ITB and BMT between baseline and months 6
Time Frame: baseline, ITB test (only ITB arm), second assessment (only BMT arm), week 6 (only ITB arm), month 3, month 6
Population: Intent to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ITB Therapy | Best Medical Treatment (BMT)
Number analyzed (Participants) | 31 | 29
Participants
  Baseline : general practitioner | 14 | 8
  Baseline : neurologist | 4 | 8
  Baseline : nurse (hospital setting) | 1 | 0
  Baseline : nurse (home care) | 0 | 1
  Baseline : orthopedic surgeon | 3 | 0
  Baseline : other | 10 | 13
  ITB test:general practitioner | 1 | NA — ITB test visit is not applicable for the BMT arm
  ITB test: neurologist | 1 | NA — ITB test visit is not applicable for the BMT arm
  ITB test :other | 3 | NA — ITB test visit is not applicable for the BMT arm
  Second Assessment: general practitioner | NA — Second assessemnt visit is not applicable for the ITB arm | 5
  Second Assessment: neurologist | NA — Second assessemnt visit is not applicable for the ITB arm | 1
  Second Assessment: nurse (home care) | NA — Second assessemnt visit is not applicable for the ITB arm | 1
  Second Assessment: other | NA — Second assessemnt visit is not applicable for the ITB arm | 4
  week 6: general practitioner | 4 | NA — week 6 visit is not applicable for the BMT arm
  week 6: nurse (hospital setting) | 2 | NA — week 6 visit is not applicable for the BMT arm
  week 6: other | 2 | NA — week 6 visit is not applicable for the BMT arm
  month 3: general practitioner | 7 | 8
  month 3: neurologist | 1 | 3
  month 3: other | 6 | 9
  month 6: general practitioner | 8 | 7
  month 6: neurologist | 3 | 2
  month 6: other | 8 | 11

ADVERSE EVENTS:
Time Frame: From ITB test (for ITB arm) and randomization (for BMT arm) untill month 6 follow-up visit
Description: Safety analyses were performed on a modified ITT (intent to treat) patient set: all patients were analyzed as treated; ITB-I included only implated patients. BMT+ITB-NI included also patients randomized to ITB, but not implanted.
Groups:
- ITB-I: Patients implanted with intrathecal baclofen pump
- BMT+ITB-NI: Patients randomized to BMT plus patients randomized to ITB but not implanted (treated with one or a combination oral antispastic medication)
Arm/Group | ITB-I | BMT+ITB-NI
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/35
Serious Adverse Events (participants affected / at risk) | 12/25 | 10/35
Other Adverse Events (participants affected / at risk) | 23/25 | 21/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITB-I (N=25) | BMT+ITB-NI (N=35)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (5)
Implant site infection (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (3)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 2 (2) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Implant site effusion (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITB-I (N=25) | BMT+ITB-NI (N=35)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Implant site pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 4 (4) | 3 (3)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chronic fatigue syndrome (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Implant site reaction (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (10) | 3 (4)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Residual urine volume increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hypotonia (Nervous system disorders) | 3 (3) | 0 (0)
Muscle spasticity (Nervous system disorders) | 2 (2) | 3 (3)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Sedation (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 3 (4)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Listless (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days